CLINICAL TRIAL: NCT07338734
Title: Fluid Balance During Early Hours of Acute Kidney Injury in Critically Ill Patients
Brief Title: Fluid Balance in Acute Kidney Injury in Critically Ill Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Engy Bassam Gayel Sayed, Resident at Internal Medicine Department, Assiut University, Assiut University
Other Study IDs: Fluid Balance in AKI
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Fluid Balance; Acute Kidney Injury; Critically Ill Acute Kidney Injury; Critically Ill
Keywords: Fluid Balance; acute kidney injury; AKI; critically ill; KDIGO criteria
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This prospective observational cohort study evaluates if fluid balance in the first 48 hours of ICU admission is linked to acute kidney injury (AKI) in critically ill adults. Patients without AKI at entry will have fluids tracked hourly via charts, weights, and labs to assess AKI risk by KDIGO criteria within 7 days. Findings may guide better fluid management to lower AKI rates.

DETAILED DESCRIPTION:
This prospective observational cohort study at Assiut University Hospital ICU investigates the association between fluid balance in the first 48 hours of admission and acute kidney injury (AKI) development. Critically ill adults (≥18 years) without AKI at baseline will undergo routine monitoring: hourly fluid intake/output (IV fluids, blood products, urine, drains, insensible losses), daily weights, serial labs (SCr, BUN, electrolytes, albumin, CRP), and clinical/hemodynamic assessments. AKI is defined/staged by KDIGO criteria within 7 days. Sample size is 120 (Epi-Info calculated, 38.4% expected AKI incidence). Data analysis will examine if positive/negative balances predict AKI incidence, severity, RRT need, ICU stay, and 28-day mortality, using AKI-FB risk score. No interventions; standard care only.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older admitted to the ICU.
* Patients with no AKI at ICU admission.
* AKI secondary to (prerenal cause-renal and post renal with manifestation of hypovolemia)-postoperative settings-On top of CKD up to Stage 111b-Compansated heart failure with indication of fluid therapy

Exclusion Criteria:

* Patients with pre-existing end-stage renal disease requiring dialysis.
* Patients with known chronic kidney disease stage 4 or higher.
* ICU readmissions during the same hospitalization.
* Patients who received renal replacement therapy before ICU admission
* Patients with AKI with manifestation of over load as pulmonary edema- pulmonary embolism-Acute decompensated heart failure

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years or older admitted to the intensive care unit (ICU) at Assiut University Hospital without acute kidney injury (AKI) at admission. Eligible cases include prerenal, renal, postrenal AKI with hypovolemia; postoperative; CKD up to stage IIIb; compensated heart failure needing fluids.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Acute Kidney Injury (AKI) | Within 7 days after ICU admission
  Development of AKI defined by KDIGO criteria (increase in serum creatinine by ≥0.3 mg/dL within 48 hours or ≥1.5 times baseline within 7 days, or urine output <0.5 mL/kg/h for 6 hours).

SECONDARY OUTCOMES:
AKI Stage by KDIGO Criteria | Within 7 days after ICU admission
  Worst stage of AKI (Stage 1: SCr 1.5-2.9x baseline or UO <0.5 mL/kg/h ≥6h; Stage 2: SCr 3-5.9x or UO <0.5 mL/kg/h ≥12h; Stage 3: SCr ≥6x or ≥4.0 mg/dL or RIFLE F/ESRD, UO <0.3 mL/kg/h ≥24h or anuria ≥12h).